CLINICAL TRIAL: NCT05003193
Title: The Effect of Pedometer Assisted Walking on Physical Activity Level and Metabolic Parameters in Patients With Renal Transplantation
Brief Title: The Effect of Walking in Kidney Transplant Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, FATMA DEMIR KORKMAZ, Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: fatma.demir1
Record Dates: First submitted 2021-03-30; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Kidney Transplant; Complications; Cardiac Disease
Keywords: transplantation; exersize; heart diseases; kidney; nursing care
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using a pedometer (Experimental): The pedometer will be given to the intervention group to evaluate the activity level and to encourage a walk , it will be said that their goal is to take 2000 steps in 20 minutes a day after discharge. Patients will be asked to carry the pedometer during physical activity, and to write down the number of steps they take in 20 minutes on the form given to them for 90 days.
  Interventions: Device: pedometer
- Not using a pedometer (No Intervention): The control group will not be given a pedometer.Patients in the control group will only be instructed to do physical activity every day and will be asked to record the minutes of physical activity they do for 90 days.

INTERVENTIONS:
Device: pedometer — 2000 steps per day in 20 minutes for 90 days, guided by a pedometer after a kidney transplantation
  Arms: Using a pedometer

SUMMARY:
Cardiovascular diseases are among the most common causes of death in kidney transplant patients. Physical activity is of great importance in preventing cardiovascular diseases after transplantation. Although regular physical activity is recommended in international guidelines to prevent post-transplant mortality and morbidity in kidney transplant patients, studies have shown that patients do not follow regular physical activity instructions.The aim of our project is to examine the effect of pedometer-assisted physical activity on metabolic parameters after kidney transplantation.

DETAILED DESCRIPTION:
Patients with kidney transplant surgery will be randomized to the intervention (n: 34) and control groups (n: 34), respectively, according to the transplant surgery date. Intervention and Control groups will be given the same training on the importance of physical activity during discharge training. The pedometer will be given to the intervention group to evaluate the activity level, and it will be said that their goal is to take 2000 steps in 20 minutes a day after discharge. Patients will be asked to carry the pedometer during physical activity, and to write down the number of steps they take in 20 minutes on the form given to them for 90 days. Patients in the control group will only be advised to do physical activity every day and will be asked to record the minutes of physical activity they do for 90 days. Metabolic parameters of the patients in the intervention and control groups will be examined at the end of the 4th and 12th months. These parameters are blood pressure, body mass index, complete blood count (hemoglobin, leukocyte, thrombocyte), blood glucose, sodium, potassium, calcium, liver enzymes, serum creatinine, total and indirect bilirubin, albumin and total cholesterol levels.

ELIGIBILITY:
Inclusion Criteria: • Over the age of 18 and under the age of 65,

* Kidney transplantation at the center where the study was conducted between the research dates,
* There is no activity restriction recommendation by the physician,
* Patients who agree to participate in the study.

Exclusion Criteria:

* Multiple organ transplantation at the same time,
* Death or graft loss/rejection in the hospital before discharge,
* Patients with physical activity restrictions by the physician,
* Patients who are re-hospitalized within the first 3 months after discharge

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Change from Baseline Blood Pressure at 4 months after discharge
  mmHg
Blood Pressure | Change from Baseline Blood Pressure at 12 months after discharge
  mmHg
Body Mass Index (BMI) | Change from Baseline BMI at 4 months after discharge
  BMI is weight in kilograms divided by height in meters squared. Formula: weight (kg) / [height (m)]2
Body Mass Index (BMI) | Change from Baseline BMI at 12 months after discharge
  BMI is weight in kilograms divided by height in meters squared. Formula: weight (kg) / [height (m)]2
Hemoglobin | Change from Baseline Hemoglobin at 4 months after discharge
  g/dL
Hemoglobin | Change from Baseline Hemoglobin at 12 months after discharge
  g/dL
Leukocyte | Change from Baseline Leukocyte at 4 months after discharge
  10^3/µL
Leukocyte | Change from Baseline Leukocyte at 12 months after discharge
  10^3/µL
Thrombocyte | Change from Baseline Thrombocyte at 4 months after discharge
  10^3/µL
Thrombocyte | Change from Baseline Thrombocyte at 12 months after discharge
  10^3/µL
Blood Glucose | Change from Baseline Blood Glucose at 4 months after discharge
  mg/dL
Blood Glucose | Change from Baseline Blood Glucose at 12 months after discharge
  mg/dL
Sodium | Change from Baseline Sodium at 4 months after discharge
  mEq/L
Sodium | Change from Baseline Sodium at 12 months after discharge
  mEq/L
Potassium | Change from Baseline Sodium at 4 months after discharge
  mEq/L
Potassium | Change from Baseline Sodium at 12 months after discharge
  mEq/L
Calcium | Change from Baseline Sodium at 4 months after discharge
  mEq/L
Calcium | Change from Baseline Sodium at 12 months after discharge
  mEq/L
Serum Creatinine | Change from Baseline Sodium at 4 months after discharge
  mg/dL
Serum Creatinine | Change from Baseline Sodium at 12 months after discharge
  mg/dL
Total Bilirubin | Change from Baseline Sodium at 4 months after discharge
  mg/dL
Total Bilirubin | Change from Baseline Sodium at 12 months after discharge
  mg/dL
Indirect Bilirubin | Change from Baseline Sodium at 4 months after discharge
  mg/dL
Indirect Bilirubin | Change from Baseline Sodium at 12 months after discharge
  mg/dL
High-density lipoprotein (HDL) cholesterol | Change from Baseline Sodium at 4 months after discharge
  mg/dL
High-density lipoprotein (HDL) cholesterol | Change from Baseline Sodium at 12 months after discharge
  mg/dL
Low-density lipoprotein (LDL) cholesterol | Change from Baseline Sodium at 4 months after discharge
  mg/dL
Low-density lipoprotein (LDL) cholesterol | Change from Baseline Sodium at 12 months after discharge
  mg/dL
Aspartate Aminotransferase | Change from Baseline Sodium at 4 months after discharge
  U/L
Aspartate Aminotransferase | Change from Baseline Sodium at 12 months after discharge
  U/L
Alanine aminotransferase | Change from Baseline Sodium at 4 months after discharge
  U/L
Alanine aminotransferase | Change from Baseline Sodium at 12 months after discharge
  U/L
Alkaline Phosphatase | Change from Baseline Sodium at 4 months after discharge
  U/L
Alkaline Phosphatase | Change from Baseline Sodium at 12 months after discharge
  U/L
Triglyceride | Change from Baseline Sodium at 4 months after discharge
  mg/dL
Triglyceride | Change from Baseline Sodium at 12 months after discharge
  mg/dL
Total Cholesterol | Change from Baseline Sodium at 4 months after discharge
  mg/dL
Total Cholesterol | Change from Baseline Sodium at 12 months after discharge
  mg/dL
Albumin | Change from Baseline Sodium at 4 months after discharge
  g/dL
Albumin | Change from Baseline Sodium at 12 months after discharge
  g/dL
glucose in urine | Change from Baseline Sodium at 4 months after discharge
  mg/dL
glucose in urine | Change from Baseline Sodium at 12 months after discharge
  mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Fatma DEMIR KORKMAZ, Professor, Principal Investigator — Ege University Faculty of Nursing 35000, Izmir, Turkey
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Zelle DM, Kok T, Dontje ML, Danchell EI, Navis G, van Son WJ, Bakker SJ, Corpeleijn E. The role of diet and physical activity in post-transplant weight gain after renal transplantation. Clin Transplant. 2013 Jul-Aug;27(4):E484-90. doi: 10.1111/ctr.12149. Epub 2013 Jun 13. PMID 23758229
- [Background] Zelle DM, Corpeleijn E, Klaassen G, Schutte E, Navis G, Bakker SJ. Fear of Movement and Low Self-Efficacy Are Important Barriers in Physical Activity after Renal Transplantation. PLoS One. 2016 Feb 4;11(2):e0147609. doi: 10.1371/journal.pone.0147609. eCollection 2016. PMID 26844883
- [Background] Lorenz EC, Amer H, Dean PG, Stegall MD, Cosio FG, Cheville AL. Adherence to a pedometer-based physical activity intervention following kidney transplant and impact on metabolic parameters. Clin Transplant. 2015 Jun;29(6):560-8. doi: 10.1111/ctr.12553. Epub 2015 May 26. PMID 25845820
- [Background] Gustaw T, Schoo E, Barbalinardo C, Rodrigues N, Zameni Y, Motta VN, Mathur S, Janaudis-Ferreira T. Physical activity in solid organ transplant recipients: Participation, predictors, barriers, and facilitators. Clin Transplant. 2017 Apr;31(4). doi: 10.1111/ctr.12929. Epub 2017 Mar 14. PMID 28185297
- [Background] Aakhus S, Dahl K, Wideroe TE. Cardiovascular disease in stable renal transplant patients in Norway: morbidity and mortality during a 5-yr follow-up. Clin Transplant. 2004 Oct;18(5):596-604. doi: 10.1111/j.1399-0012.2004.00235.x. PMID 15344967
- [Background] Ojo AO. Cardiovascular complications after renal transplantation and their prevention. Transplantation. 2006 Sep 15;82(5):603-11. doi: 10.1097/01.tp.0000235527.81917.fe. PMID 16969281
- [Background] Berben L, Engberg SJ, Rossmeissl A, Gordon EJ, Kugler C, Schmidt-Trucksass A, Klem ML, Sereika SM, De Simone P, Dobbels F, De Geest SM; B-SERIOUS consortium. Correlates and Outcomes of Low Physical Activity Posttransplant: A Systematic Review and Meta-Analysis. Transplantation. 2019 Apr;103(4):679-688. doi: 10.1097/TP.0000000000002543. PMID 30461720
- [Background] Dontje ML, de Greef MH, Krijnen WP, Corpeleijn E, Kok T, Bakker SJ, Stolk RP, van der Schans CP. Longitudinal measurement of physical activity following kidney transplantation. Clin Transplant. 2014 Apr;28(4):394-402. doi: 10.1111/ctr.12325. Epub 2014 Mar 17. PMID 24635476
- [Background] Gordon EJ, Prohaska TR, Gallant MP, Sehgal AR, Strogatz D, Yucel R, Conti D, Siminoff LA. Longitudinal analysis of physical activity, fluid intake, and graft function among kidney transplant recipients. Transpl Int. 2009 Oct;22(10):990-8. doi: 10.1111/j.1432-2277.2009.00917.x. Epub 2009 Jul 10. PMID 19619168
- [Background] Hawkins MS, Sevick MA, Richardson CR, Fried LF, Arena VC, Kriska AM. Association between physical activity and kidney function: National Health and Nutrition Examination Survey. Med Sci Sports Exerc. 2011 Aug;43(8):1457-64. doi: 10.1249/MSS.0b013e31820c0130. PMID 21200336
- [Background] Svensson M, Jardine A, Fellstrom B, Holdaas H. Prevention of cardiovascular disease after renal transplantation. Curr Opin Organ Transplant. 2012 Aug;17(4):393-400. doi: 10.1097/MOT.0b013e3283560a3b. PMID 22790074
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C; American College of Sports Medicine; American Heart Association. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1094-105. doi: 10.1161/CIRCULATIONAHA.107.185650. Epub 2007 Aug 1. PMID 17671236
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Transplant Work Group. KDIGO clinical practice guideline for the care of kidney transplant recipients. Am J Transplant. 2009 Nov;9 Suppl 3:S1-155. doi: 10.1111/j.1600-6143.2009.02834.x. PMID 19845597